CLINICAL TRIAL: NCT07298473
Title: Conquer-AF Protocol for Redo Ablation Procedures in Recurrent Paroxysmal and Persistent Atrial Fibrillation Using the Sphere-9 Catheter and Affera Ablation System (Conquer-AF)
Acronym: Conquer-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT25005
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF); Persistent Atrial Fibrillation; Paroxysmal Atrial Fibrillation (PAF)
Keywords: Sphere-9 Catheter; Affera Ablation System; Affera Mapping System; Pulsed Field Ablation (PFA); Radiofrequency Ablation (RFA); Dual-Energy Ablation; Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation; Redo Ablation; Repeat Ablation; Electrophysiology Mapping; 3D Cardiac Mapping; Left Atrial Ablation; Redo AF Ablation; Repeat Ablation Procedures
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-center, single-arm study in which all enrolled participants undergo a redo atrial fibrillation ablation using the Sphere-9 Catheter and Affera Ablation System. There is no randomization or control groups.
  All subjects who have the Sphere-9™ Catheter inserted into the vasculature are included in the Primary Analysis Group. Subjects who exit the study prior to catheter insertion are classified as non-treated and are not included in the primary analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single Arm: Redo AF Ablation with Sphere-9 Catheter (Experimental): Participants undergo a redo atrial fibrillation ablation using the Sphere-9 Catheter and the Affera Ablation System per study protocol. All subjects receive the same intervention with no control or comparator arm.
  Interventions: Device: Sphere-9 Catheter Ablation

INTERVENTIONS:
Device: Sphere-9 Catheter Ablation — Redo atrial fibrillation ablation performed using the Sphere-9 Catheter in conjunction with the Affera Ablation System and Affera Mapping System. The intervention delivers radiofrequency and pulsed field energy according to the study protocol for treatment of recurrent paroxysmal or persistent AF. All participants receive this device-based ablation procedure.
  Other Names: Affera Ablation System; Affera Mapping System

SUMMARY:
Conquer-AF is a prospective, multi-center, interventional, non-randomized clinical study that will enroll up to 400 subjects at up to 30 sites across the United States, Europe, and Australia.

Subjects diagnosed with symptomatic recurrent paroxysmal or persistent atrial fibrillation after a single prior ablation procedure will be enrolled in this study. Each subject will undergo a study index redo ablation procedure using the Sphere-9 Catheter and Affera Ablation System and will be followed for 12 months. The expected total study duration (from time of first enrollment to the exit of last enrolled subject) is approximately 2 years.

DETAILED DESCRIPTION:
The Conquer-AF study is a prospective, multi-center, interventional, non-randomized clinical study to evaluate the safety and effectiveness of the Sphere-9 Catheter and Affera Ablation System, when used in conjunction with the Affera Mapping System or Affera Integrated Mapping System, in patients undergoing redo ablation for symptomatic recurrent paroxysmal or persistent atrial fibrillation following a single prior ablation procedure.

This study will enroll up to 400 subjects diagnosed with symptomatic recurrent PAF and PsAF and will be conducted at up to 30 study sites located across the United States, Europe, and Australia. No single site may enroll more than 60 (with no more than 37 in either cohort) subjects to ensure a reasonable distribution of subjects across sites.

Adult subjects with symptomatic recurrent PAF and PsAF will undergo a study index redo ablation procedure with the Sphere-9 Catheter and Affera Ablation System. Following the study index redo ablation procedure and hospital discharge, all study subjects will be followed at 7 days, 3 months, 6 months, and 12 months post-procedure. Subjects will be exited from the study at the conclusion of the 12-month follow-up visit and associated 24-hour Holter. The expected total study duration is approximately 2 years, representing approximately 12 months of enrollment and 12 months of subject follow-up. Treated subjects will not be replaced with newly enrolled subjects upon early study exit.

ELIGIBILITY:
Inclusion Criteria:

* 1. History of a single AF ablation procedure for PAF or PsAF within 3 years prior to enrollment 2. Documented evidence of symptomatic AF, AT or AFL recurrence at least 90 days after subject's de novo ablation procedure, as demonstrated by:

  * A physicians' note indicating at least 1 symptomatic AF, AT, or AFL episode occurring within 12 months prior to the enrollment; and
  * At least 1 electrocardiographically documented episode of AF, AT, or AFL within 12 months prior to enrollment 3. Adults who are ≥18 years of age on the day of enrollment 4. Willing and able to comply with all study requirements and provide informed consent

Exclusion Criteria:

* 1. Continuous AF lasting for 12 months or longer 2. LA anteroposterior >55 mm (by MRI, CT, or TTE), or if LA diameter not available, non-index volume >100 mL for PsAF subjects; OR LA anteroposterior >50 mm (by MRI, CT, or TTE), or if LA diameter not available, non-index volume >95 mL for PAF subjects 3. Previous left atrial percutaneous interventions including left atrial appendage occlusion and septal closure devices 4. Planned left atrial appendage (LAA) closure procedure, cardiac transplantation or implant of a permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardiac defibrillator (with or without biventricular pacing function) for any time during the follow-up period 5. More than 1 previous AF ablation procedure 6. Any prior surgical ablation procedure 7. Patient who is not on oral anticoagulation therapy for at least 3 weeks prior to the ablation procedure 8. Contraindication to or unwillingness to use systemic anticoagulation 9. Severe thrombocytosis, thrombocytopenia, or any bleeding or clotting disorder 10. Presence of a permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardiac defibrillator (with or without biventricular pacing function) 11. Presence of any pulmonary vein stents 12. Known pre-existing pulmonary vein stenosis 13. Pre-existing hemidiaphragmatic paralysis 14. Prior valvular (surgical or percutaneous) procedure including prosthetic, bioprosthetic, valve replacement, valve repair or valvuloplasty, or any prior atriotomy 15. Moderate to severe mitral valve or aortic stenosis 16. Moderate to severe mitral regurgitation (i.e., 3+ or 4+ MR) 17. Any cardiac surgery, myocardial infarction, PCI/PTCA or coronary artery stenting which occurred within the 3 months preceding the consent date 18. NYHA Class III or IV congestive heart failure 19. Documented left ventricular ejection fraction (LVEF) ≤40%, measured by acceptable cardiac testing (e.g., TTE) 20. Unstable angina 21. Severe lung disease, primary pulmonary hypertension, or any lung disease requiring supplemental oxygen 22. Rheumatic heart disease 23. Significant restrictive or obstructive pulmonary disease or chronic respiratory condition 24. Presence of left atrial thrombus on imaging 25. Active systemic infection or sepsis 26. Hypertrophic cardiomyopathy 27. Amyloid heart disease 28. Diagnosed atrial myxoma 29. Known reversible causes of AF (e.g., uncontrolled hyperthyroidism, severe untreated obstructive sleep apnea, acute alcohol toxicity or other reversible or non-cardiac cause) 30. Any cerebral ischemic event (strokes or TIAs) which occurred within the preceding 6 months of the consent date through the date of study index redo ablation procedure 31. Carotid stenting or endarterectomy 32. Thromboembolic event within the past 6 months or evidence of intracardiac thrombus at the time of the procedure 33. Body mass index > 40 kg/m2 34. Any woman known to be pregnant or breastfeeding, or any woman of childbearing potential who is not on a reliable form of birth regulation method or abstinence* 35. Patient with life expectancy that makes it unlikely 12 months of follow-up will be completed 36. Current or anticipated participation in any other clinical study of a drug, device or biologic during the duration of the study not pre-approved by Medtronic 37. Renal insufficiency with an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2, or any history of renal failure requiring dialysis or renal transplant 38. Presence of intramural thrombus, tumor, or other abnormality that precludes vascular access, catheter introduction, or manipulation 39. Presence of an inferior vena cava (IVC) filter (e.g., Greenfield or similar) that would preclude safe transfemoral venous access, catheter passage, or sheath manipulation.

  40. Known drug or alcohol dependency 41. Significant congenital anomaly or medical problem that would, in the opinion of the investigator, preclude enrollment, follow-up compliance, or the scientific integrity of the study

  *Women who are of child-bearing potential must undergo a pregnancy test after consent and prior to the study index redo ablation procedure, as allowed according to local regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-03-29 (Estimated); Study Completion 2028-03-29 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: Number of Participants With Treatment Success. | 12-months post-redo ablation procedure
  Treatment success is defined to be freedom from treatment failure. The study requires 24-hour Holter monitoring at 6 and 12 months, weekly and symptomatic patient activated TTM transmissions through 12 months, and 12-lead ECGs or TTMs at all follow up visits. Treatment failure is defined as any of the following components:
  * Inability to successfully complete the study index redo ablation procedure utilizing the Sphere-9 Catheter and Affera Ablation System exclusively
  * Documented AF/AT/AFL after the 90-day post-ablation blanking period
  * Any subsequent catheter or surgical ablation, for recurrent AF/AT/AFL including repeat redo ablation at any time during the study
  * Direct current or pharmacological cardioversion for AF/AT/AFL recurrences after the 90-day blanking period (See section 9.11)
  * Use of a Class I or III AAD at a higher daily dose than the pre-ablation maximum dose after the 90-day blanking period and on or before day 365.
  * Initiation of a new Class I or III AAD after t
Safety: Number of Participants With at Least One Primary Safety Event | 6-months post-redo ablation procedure
  Primary safety events include:
  * 7 days of post-ablation: AKI requiring dialysis, new hospitalization >48 hours, or prolongation of hospitalization >48 hours beyond expected discharge, Death, Heart block requiring pacemaker, Major bleeding requiring transfusion, MI, Permanent phrenic nerve paralysis, Pulmonary edema, Severe pericarditis, Significant pericardial effusion/tamponade, Stroke/CVA, Systemic/pulmonary embolism requiring intervention, TIA, Vagal nerve injury resulting in esophageal dysmotility or gastroparesis, Vascular access complications requiring intervention, Any Sphere-9 Catheter or Affera Mapping & Ablation System device- or procedure-related cardiovascular and/or pulmonary AE that prolongs or requires hospitalization >48 hours (excl recurrent AF/AT/AFL)
  * 3 months post-ablation: Atrioesophageal fistula/esophago-pericardial fistula, Esophageal perforation (procedure & Sphere-9 Catheter related)
  * 6 months post-ablation: Pulmonary vein stenosis (≥70% diameter reduction)

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Tarakji, MD, Study Director — Medtronic

IPD SHARING:
Plan to Share IPD: No